CLINICAL TRIAL: NCT04621110
Title: Intranasal Dexmedetomidine and Fentanyl Versus Intravenous Midazolam and Ketamine in Sedation for Painful Outpatient Procedures
Brief Title: Intranasal Versus Intravenous Drug in Painful Procedure for Outpatient Oncologic Participants
Acronym: NAIVe
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Eduardo Juan Troster, Associate Professor, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dexmedetomidine4040519
Record Dates: First submitted 2020-09-29; First posted 2020-11-09 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Pediatric Cancer; Analgesia; Procedural Pain
Keywords: fentanyl; dexmedetomidine
MeSH Terms: conditions — Neoplasms; Agnosia; Pain, Procedural | interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intranasal dexmedetomidine and fentanyl (Experimental): Dexmedetomidine (precedex®) and fentanyl will be administered by intranasal routes, seeing if both sedative (dexmedetomidine) and analgesic (fentanyl) can give enough sedation for procedure
  Interventions: Drug: intranasal dexmedetomidine; Drug: intranasal fentanyl
- intravenous ketamine and midazolam (Active Comparator): ketamine (ketalar®) and midazolam intravenous will be using to compare the efficiency of intranasal drugs
  Interventions: Drug: intravenous ketamine (ketalar®); Drug: intravenous midazolam

INTERVENTIONS:
Drug: intranasal dexmedetomidine — Dexmedetomidine (precedex®) will be administered by intranasal route in 1ug/kg each dose, repeating at most 3 times to see if it can give enough sedation to painful procedure. To assess the level of sedation the study will use Ramsay sedation scale.
  Arms: intranasal dexmedetomidine and fentanyl
Drug: intranasal fentanyl — Fentanyl will be administered by intranasal route in 1,5ug/kg each dose, repeating at most 3 times to see if it can give enough pain relief for painful procedure. To assess pain control the study will use Face, Legs, Activity, Cry, Consolability scale ( FLACC)
  Arms: intranasal dexmedetomidine and fentanyl
Drug: intravenous ketamine (ketalar®) — Ketamine (ketalar®) will be administrated by intravenous route in 1mg/kg dose and the study will use this drug to compare the efficiency of intranasal drugs.
  Arms: intravenous ketamine and midazolam
Drug: intravenous midazolam — Midazolam will be administrated by intravenous route in 0,1mg/kg dose and the study will use this drug to compare the efficiency of intranasal drugs.
  Arms: intravenous ketamine and midazolam

SUMMARY:
Pain is a vital sign that depends on personal experience involving different factors such as previous sensory and emotional experience, age, spiritual and cultural aspects, that makes it harder to evaluate, especially in young children. Pain control is important to diminish the anxiety of the child and family, also this is more important in patients who require procedure and treatment that are more painful, like oncological and hematological patients. The study aims to measure if the intranasal drugs (dexmedetomidine and fentanyl) has the same outcomes when compared with intravenous drug (ketamine and midazolam), but with less side effects. The participants are patients from an oncologic outpatient, that will be submitted to cerebrospinal fluid puncture, myelogram or both will be randomized assigned to both groups. The study will compare physiological variables ( heart rate, respiratory rate and blood pressure) and sedation and pain scales to see if its work properly. The study purpose is to evaluate if intranasal drug works in the same way with less side effects comparing with the usual treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with oncohematological diseases that requires cerebrospinal fluid, myelogram or both for staging and monitoring their treatment ( leukemia, lymphoma, solid tumors and bone marrow aplasia)
* Patients who is undergoing to collect cerebrospinal fluid, myelogram or both;
* aged between two and eight years;
* absence of tumor recurrence.

Exclusion Criteria:

* Previous neurologic disease;
* Using of opioid previously;
* Neurological developmental delay

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Pain control | The FLACC scale will be measure each 2 minutes up to 30 minutes.
  Evaluate if intranasal drugs is effective for pain relief in painful procedures for paediatric oncologic and hematologic patients. To measure it will use Face, Legs, Activity, Cry, Consolability scale (FLACC). This is a scale for pain in children, and for each sign gives 0-2 point, and 0 is no pain and 7-10 intense pain
Sedation | The Ramsay scale will be measure each 2 minutes up to 30 minutes.
  Evaluate if intranasal drugs is effective for sedation in painful procedures for paediatric oncologic and hematologic patients. For access this, will be use Ramsay scale, this scale range between 1 to 6. 1 is a anxious patient and 6 sleeping patient without answer
Change in heart rate | each 2 minutes up to 30 minutes
  evaluate side effects using PALS ( paediatric advanced life support) values for ages. To evaluate this, heart rate values will be noted before the procedure, during and after that and will be evaluated if there was an increase or decrease in it, respecting a significance level of 5%.
Change in respiratory rate | each 2 minutes up to 30 minutes
  evaluate side effects using PALS ( paediatric advanced life support) values for different ages. To evaluate this, respiratory rate values will be noted before the procedure, during and after that and will be evaluated if there was an increase or decrease in it, respecting a significance level of 5%.
Change in blood pressure | each 2 minutes up to 30 minutes
  evaluate side effects using PALS ( paediatric advanced life support) values for ages. To evaluate this, blood pressure value will be noted before the procedure, during and after that and will be evaluated if there was an increase or decrease in it, respecting a significance level of 5%.

SECONDARY OUTCOMES:
Comparison if intranasal drugs has the same pain relief as intravenous drugs | each 2 minutes up to 30 minutes
  Using Face, Legs, Activity, Cry, Consolability (FLACC) to compare both arms. The FLACC is a scale for pain in children, and for each sign gives 0-2 point, and 0 is no pain and 7-10 intense pain
Comparison if intranasal drugs has the same sedation effects like intravenous drug | each 2 minutes after medication up to 30 minutes
  Using Ramsay scale to compare both arms, intranasal and intravenous drugs. The Ramsay scale range between 1 to 6. 1 is a anxious patient and 6 sleeping patient without answer effect in sedation.

CONTACTS AND LOCATIONS:
Locations (1):
- ITACI - Instituto de Tratamento do Câncer Infantil/ ICR HCFMUSP, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Manworren RC, Stinson J. Pediatric Pain Measurement, Assessment, and Evaluation. Semin Pediatr Neurol. 2016 Aug;23(3):189-200. doi: 10.1016/j.spen.2016.10.001. Epub 2016 Oct 17. PMID 27989326
- [Background] Fantacci C, Fabrizio GC, Ferrara P, Franceschi F, Chiaretti A. Intranasal drug administration for procedural sedation in children admitted to pediatric Emergency Room. Eur Rev Med Pharmacol Sci. 2018 Jan;22(1):217-222. doi: 10.26355/eurrev_201801_14120. PMID 29364490
- [Background] Li BL, Zhang N, Huang JX, Qiu QQ, Tian H, Ni J, Song XR, Yuen VM, Irwin MG. A comparison of intranasal dexmedetomidine for sedation in children administered either by atomiser or by drops. Anaesthesia. 2016 May;71(5):522-8. doi: 10.1111/anae.13407. Epub 2016 Mar 3. PMID 26936022
- [Background] Tug A, Hanci A, Turk HS, Aybey F, Isil CT, Sayin P, Oba S. Comparison of Two Different Intranasal Doses of Dexmedetomidine in Children for Magnetic Resonance Imaging Sedation. Paediatr Drugs. 2015 Dec;17(6):479-85. doi: 10.1007/s40272-015-0145-1. PMID 26323489
- [Background] Jun JH, Kim KN, Kim JY, Song SM. The effects of intranasal dexmedetomidine premedication in children: a systematic review and meta-analysis. Can J Anaesth. 2017 Sep;64(9):947-961. doi: 10.1007/s12630-017-0917-x. Epub 2017 Jun 21. PMID 28639236
- [Background] Gupta A, Dalvi NP, Tendolkar BA. Comparison between intranasal dexmedetomidine and intranasal midazolam as premedication for brain magnetic resonance imaging in pediatric patients: A prospective randomized double blind trial. J Anaesthesiol Clin Pharmacol. 2017 Apr-Jun;33(2):236-240. doi: 10.4103/joacp.JOACP_204_16. PMID 28781452
- [Background] Chatrath V, Kumar R, Sachdeva U, Thakur M. Intranasal Fentanyl, Midazolam and Dexmedetomidine as Premedication in Pediatric Patients. Anesth Essays Res. 2018 Jul-Sep;12(3):748-753. doi: 10.4103/aer.AER_97_18. PMID 30283188
- [Background] Kleinman ME, Chameides L, Schexnayder SM, Samson RA, Hazinski MF, Atkins DL, Berg MD, de Caen AR, Fink EL, Freid EB, Hickey RW, Marino BS, Nadkarni VM, Proctor LT, Qureshi FA, Sartorelli K, Topjian A, van der Jagt EW, Zaritsky AL. Part 14: pediatric advanced life support: 2010 American Heart Association Guidelines for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2010 Nov 2;122(18 Suppl 3):S876-908. doi: 10.1161/CIRCULATIONAHA.110.971101. No abstract available. PMID 20956230